CLINICAL TRIAL: NCT03402009
Title: Assisting University Students Self-Manage Stress: Comparison of Mindfulness Meditation Tools
Brief Title: Comparison of Mindfulness Meditation Tools For College Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Blair Johnson, BoT Distinguished Professor of Psychological Sciences, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H17-224
Record Dates: First submitted 2017-12-06; First posted 2018-01-17 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Stress; Anxiety
Keywords: meditation; Mindfulness; stress; anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Amyloid Precursor Protein Secretases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): independent meditation using web-based tools, apps, and EEG neurofeedback
  Interventions: Behavioral: Apps; Behavioral: EEG neurofeedback
- Active Control (Active Comparator): independent meditation using web-based tools and apps
  Interventions: Behavioral: Apps

INTERVENTIONS:
Behavioral: Apps — Apps and weblinks to coach self-guided meditation.
Behavioral: EEG neurofeedback — Device provides feedback based on EEG readings.
  Arms: Experimental

SUMMARY:
The purpose of this study is to determine what tools best assist university students develop a personal meditation practice to self-manage stress. The two treatment conditions are 1) independent meditation using web-based tools and apps, and 2) independent meditation using web-based tools, apps and EEG-based neurofeedback. Outcomes of interest include acceptability, adherence, changes in mental health (i.e., anxiety, stress), physical health (i.e., sleep, inflammation), resilience, and level of commitment to further practice. Factors related to self-regulation (i.e., interoceptive awareness, self-esteem) will also be assessed as potential outcome moderators.

DETAILED DESCRIPTION:
Investigators will conduct a randomized controlled trial to evaluate strategies for assisting students develop a personal meditation practice. All participants will attend a mindfulness orientation, then begin the four-week intervention. During the intervention period, the treatment group will practice EEG-neurofeedback-assisted meditation using the Muse device (Interaxon) at least eight times over the four-week intervention period, and also practice mindfulness meditation on their own using their choice of tools (e.g., apps, weblinks, breath). The active control group will mirror the treatment group but will not have access to the EEG-neurofeedback device.

After a sufficient number of students register for the study who meet eligibility requirements, they will be provided with an option to enroll online in the first wave of the study, if their schedule allows, or be placed on a waitlist. Subsequent waves will take place throughout the semester(s) to accommodate additional participants. Enrolled participants will be asked to complete the pre-workshop questionnaire packet online, and attend an orientation session. During the orientation session, participants will first sign a consent form, provide a baseline saliva sample, then learn the basic technique of mindfulness meditation with an experienced meditation instructor. The orientation will also briefly explain the potential benefits of meditation from a scientific perspective, and emphasize the importance of establishing a daily practice, with the mindset that even one minute counts. Participants will then be asked to meditate for 3 minutes wearing the EEG device in order to get a baseline EEG reading. Following the orientation workshop, participants will be randomly assigned and notified via email into either the active control or treatment group along with group-specific instructions, and the 4-week intervention period will commence. Upon completion of the 4-week intervention, participants will be asked to complete post-intervention questionnaires online, then provide post-test measures of saliva, EEG reading during a 3 minute meditation. Participants will be debriefed, and those in the active control group will be given the option to use the EEG-neurofeedback. Follow-up surveys will be emailed to participants at 3, 6 and 12 months to examine if participants continue their meditation practice.

ELIGIBILITY:
Inclusion Criteria:

* English literate, undergraduates and graduate students attending UConn ages 18 and above (unless they are registered with the participant pool), who agree with the initial terms, are willing to learn basic skills of mindfulness meditation, agree to practice meditating with assigned tools independently and feel able to adhere to the time commitment required for the study. Participants must not currently have a regular seated meditation practice (regular, meaning at least 1x per week).

Exclusion Criteria:

* participants unable to adhere to the commitment required for the study will be excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Depression, Anxiety, and Stress Scales-21 | 5 weeks
  (DASS-21; Lovibond & Lovibond, 1995): an abbreviated, 21-item, Likert-style scale to assess levels of distress on three subscales: depression, anxiety and stress, based on how one felt over the past week. The DASS-21 has been used in prior studies assessing the benefits of mindfulness in undergraduate students (Gallego et al., 2014). It consists of 21 items with seven items per subscale, scored on a four-point scale ranging from 0 = did not apply to me at all to 3 = applied to me very much or most of the time. The total score sums all items. Higher scores indicate higher levels of distress.

SECONDARY OUTCOMES:
Big Five personality | Baseline and 5 weeks
  Big Five personality traits (Costa & McCrae, 1992), which are openness, conscientiousness, extraversion, agreeableness, and neuroticism. These factors have been used to understand the relationship between personality and various academic behaviors. Respondents rate each item on a five-point scale from "strongly disagree" to "strongly agree." This scale been used extensively in psychology research and has demonstrated good internal consistency, test-retest reliability, and validity (Costa & McCrae, 1992).
Pittsburgh Sleep Quality Index | Baseline and 5 weeks
  Sleep quality will be assessed using the The Pittsburgh Sleep Quality Index (PSQI) (Buysse et al, 1989), a commonly used, validated and reliable measure of sleep quality.
Self-Regulation of Eating Scale | Baseline and 5 weeks
  The Self-Regulation of Eating Behavior Questionnaire (SREBQ) is a short, Likert format questionnaire comprising of two dichotomous screener questions, one directional question to bring tempting foods to mind, and five Likert-format items assessing respondents' self-regulation of eating. The five Likert-format items span a five-point scale from 'Never' to 'Always'. The SREBQ has been shown to be reliable and valid (Kliemann et al., 2016).
MINDSENS (mindfulness) | Baseline and 5 weeks
  a composite index consisting of selected items from two other mindfulness questionnaires (The Five Facet Mindfulness Questionnaire and Experiences Questionnaire) that showed the strongest response to practice.
Multidimensional Assessment of Interoceptive Awareness (MAIA) | Baseline and 5 weeks
  Interoceptive self-awareness. Interoception refers to the signaling and perception of internal bodily sensations, which we will assess using the validated Multidimensional Assessment of Interoceptive Awareness (MAIA) (Mehling et. al., 2009 and 2012). The MAIA is a relatively new scale, with good validity and reliability in studies to date (Mehling et. al., 2009 and 2012; Bornemann et. Al., 2014).
Emotion Regulation Questionnaire (ERQ) | Baseline and 5 weeks
  ) (Gross & John, 2003). The ERQ assesses two specific emotion regulation strategies, suppression and reappraisal. The ERQ comprises 10 items (5 for suppression and 5 for reappraisal) rated from 1 (never do this) to 7 (always do this). The ERQ has demonstrated strong psychometric properties (Spaapen et al., 2014).
Experiences Questionnaire (decentering) | Baseline and 5 weeks
  Decentering, a specific component of mindfulness related to learning how to separate from one's own thoughts and emotions, will be assessed with the Experiences Questionnaire (Fresco 2007).
Rosenberg (1965) self-esteem scale (RSES) | Baseline and 5 weeks
  a self-esteem measure widely used in social-science research, with a scale of 0 (low) to 30 (high). It is a ten-item Likert-type scale with items answered on a four-point scale-from strongly agree to strongly disagree. It has been used extensively in research and has demonstrated good internal consistency, test-retest reliability, and validity.
Inflammatory cytokines (i.e., C-reactive protein, IL-6, and TNF-α) | Baseline and 5 weeks
  Saliva samples will be obtained in-person, during pre- and post- assessments. Saliva samples will be stored for analysis to be performed at a later date, pending funding. Future analysis on saliva will be limited to assays on stress and health-related biomarkers and inflammatory cytokines (i.e., C-reactive protein, IL-6, and TNF-α). The "passive drool" method will be used to collect saliva samples, as described in Walsh et al., 2016.
State-Trait Anxiety Inventory (STAI) | Baseline and 5 weeks
  Inventory aimed to measure one's awareness of their levels of both state and trait anxiety.
Connor-Davidson Resilience Scale (CD-RISC; Connor & Davidson, 2003) | Baseline and 5 weeks
  The CD-RISC is a 25-item scale that measures the ability to cope with stress and adversity. Items include: "I am able to adapt when changes occur," "I tend to bounce back after illness, injury, or other hardships," and "I am able to handle unpleasant or painful feelings like sadness, fear, and anger." Respondents rate items on a scale from 0 ("not true at all") to 4 ("true nearly all the time"). A preliminary study of the psychometric properties of the CD-RISC in general population and patient samples showed it to have adequate internal consistency, test-retest reliability, and convergent and divergent validity (Connor & Davidson, 2003). This measure has been used in studies that assess resilience across the lifespan (Campbell-Sills et al., 2006).
Perceived Stress Scale-4 (PSS4) | Baseline and 5 weeks
  (PSS4) is an abbreviated, 4-item Likert format scale designed to measure the degree to which situations in one's life are appraised as stressful (Cohen et al., 1983). The PSS is a validated, publicly available, and widely used psychological instrument for measuring stress. Each item asks the participant to appraise his or her feelings and thoughts using a 5-point Likert scale (0 = never, 4 = very often)

OTHER OUTCOMES:
Long-term Follow-up Survey | 1, 6, and 12 months following completion of the satisfaction follow-up
  Simple 2 question survey will ask participants if they are still meditating, and if so, what tools they are using for assistance.
Satisfaction with Mindfulness Tools | 5 weeks
  After the completion of the 4-week trial, an 18-item instrument will be used to solicit participants' satisfaction with the meditation tools, as well as their feelings toward their meditation practice as a result of the intervention (i.e.,. confidence in ability, motivation to continue, and perceived benefits). The instrument was developed for this study and asks questions about perceived benefits of mindfulness meditation and intentions to continue practicing in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Blair T. Johnson, PhD, Principal Investigator — University of Connecticut - BOT Distinguished Professor of Psychological Sciences
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for primary and secondary outcome measures will be made available upon request.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available after results have been published.
Access Criteria: Data access requests will be reviewed and requestors will be required to sign a Data Access Agreement